CLINICAL TRIAL: NCT00009880
Title: Non-Operative Therapy Of Local-Regional Carcinoma Of The Esophagus: A Randomizd Phase II Study Of Two Paclitaxel-Based Chemoradiotherapy Regimens
Brief Title: Combination Chemotherapy Plus Radiation Therapy With or Without Fluorouracil in Treating Patients With Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-0113; CDR0000068420
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2004-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the stomach; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Filgrastim; Cisplatin; Fluorouracil; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: fluorouracil
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of combination chemotherapy plus radiation therapy with and without fluorouracil in treating patients who have cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival and failure patterns in patients with previously untreated carcinoma of the esophagus or gastroesophageal junction treated with cisplatin, paclitaxel, and concurrent radiotherapy with or without fluorouracil.
* Compare the tolerance of these regimens by these patients.
* Compare the overall quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to percentage of weight loss (less than 10% vs 10% or more), disease histology (adenocarcinoma vs squamous cell carcinoma), and lesion size (no more than 5 cm vs more than 5 cm). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive induction chemotherapy comprising fluorouracil IV continuously over 24 hours and cisplatin IV over 1 hour on days 1-5, paclitaxel IV continuously over 24 hours on day 1, and filgrastim (G-CSF) subcutaneously daily on days 6-15. Treatment repeats every 4 weeks for up to 2 courses. Patients with stable or responsive disease after the first course of induction therapy receive a second course of therapy. Patients with local disease progression after the first course proceed to chemoradiotherapy.

Beginning on day 29 of the last course of induction chemotherapy, patients undergo radiotherapy 5 days a week for 5.5 weeks. Patients also receive fluorouracil IV continuously over 24 hours on days 1-5, 8-12, 15-19, 22-26, and 29-33, and paclitaxel IV over 3 hours on days 1, 8, 15, 22, and 29.

* Arm II: Patients receive induction chemotherapy comprising cisplatin IV and paclitaxel IV over 3 hours on day 1. Treatment continues every 3 weeks for 2 courses as in arm I.

Beginning on day 29 of the last course of induction chemotherapy, patients undergo radiotherapy as in arm I. Patients also receive cisplatin IV on days 1, 8, 15, 22, 29, and 36, and paclitaxel IV continuously over 96 hours on days 1-4, 8-11, 15-18, 22-25, 29-32, and 36-39.

Quality of life is assessed at baseline, within 1 week after radiotherapy, at 6 weeks after study completion, every 4 months for 1 year, every 6 months for 2 years, and then annually for 5 years.

Patients are followed within 8 weeks, every 4 months for 1 year, every 6 months for two years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 84 patients (42 per treatment arm) will be accrued for this study within 21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction

  * Stage I-III (T1, N1, M0; T2-4, N any, M0)

    * Supraclavicular or celiac lymph node involvement allowed
* Disease entirely confined to the esophagus or gastroesophageal junction and peri-esophageal soft tissue
* Cervical esophageal carcinoma allowed
* No tumor extension beyond 2 cm into stomach
* No multiple primary carcinomas of the esophagus
* No evidence of disseminated cancer
* No tracheoesophageal fistula or direct invasion into the mucosa of the trachea or major bronchi

  * Bronchoscopy with biopsy and cytology required if the primary carcinoma is less than 26 cm from the incisors or is at or above the carina by imaging study

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 65 mL/min

Cardiovascular:

* No uncontrolled heart disease
* No uncontrolled hypertension

Other:

* Total oral/enteral intake must be at least 1,700 kCal/day
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled diabetes
* No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior chest radiotherapy

Surgery:

* No prior major esophageal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (66):
- United States (66):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Esther Marie Hatton Cancer Care Center at St. Elizabeth Medical Center, Edgewood, Kentucky
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Monmouth Medical Center, Long Branch, New Jersey
  - Atlantic City Medical Center - Mainland Division, Pomona, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Akron General's McDowell Cancer Center, Akron, Ohio
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Cancer Center at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Result] Ajani JA, Winter K, Komaki R, Kelsen DP, Minsky BD, Liao Z, Bradley J, Fromm M, Hornback D, Willett CG. Phase II randomized trial of two nonoperative regimens of induction chemotherapy followed by chemoradiation in patients with localized carcinoma of the esophagus: RTOG 0113. J Clin Oncol. 2008 Oct 1;26(28):4551-6. doi: 10.1200/JCO.2008.16.6918. Epub 2008 Jun 23. PMID 18574157
- [Result] Komaki R, Winter K, Ajani J: Non-operative therapy of local-regional carcinoma of the esophagus: a randomized phase II study of two paclitaxel-based chemoradiotherapy regimens (RTOG 0113). [Abstract] The American Radium Society 89th Annual Meeting, May 5-29, 2007, Amsterdam, Netherlands. A-SS-2, 1, 2007.
- [Result] Komaki R, Winter K, Ajani A, et al.: A randomized phase II study of two paclitaxel-based chemoradiotherapy regimens for patients with the non-operative esophageal carcinoma (RTOG 0113). [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-142, S79-80, 2006.